CLINICAL TRIAL: NCT04956549
Title: Reducing African Americans' Alzheimer's Disease Risk Through Exercise-Mild Cognitive Impairment Cohort
Brief Title: Reducing African American's Alzheimer's Risk Through Exercise-Mild Cognitive Impairment (RAATE-MCI)
Acronym: RAATE-MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Robert L. Newton, Jr., Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 2020-013; R01AG067765-01 (NIH)
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Dementia of Alzheimer Type

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity (Experimental): 150 minutes of physical activity weekly
  Interventions: Behavioral: Physical activity program
- Successful Aging (Experimental): Low intensity activity program and a healthy aging educational component
  Interventions: Behavioral: Successful Aging

INTERVENTIONS:
Behavioral: Physical activity program — Supervised group sessions will be held twice per week for approximately 52 weeks. Each physical activity session will last slightly approximately 80 minutes and will consist of aerobic, strength, flexibility, and balance training. The 80 minutes of activity consists of a 5 minute warm-up, 45 minutes of aerobic training, 15 minutes of strength training, 10 minutes of balance training, and a 5 minute cool-down. The physical activity group will target 150 minutes of moderate to vigorous aerobic physical activity and two days of strength training, consistent with the current physical activity recommendations.
  Arms: Physical Activity
Behavioral: Successful Aging — The successful aging group will be based on a low-intensity activity program and a healthy aging educational component. Sessions will be approximately 60 minutes in duration and will occur once per week for the first 6 months and then every other week for the remainder 6 months of the study. The physical activities will include stretching, balance training, flexibility, relaxation, and practicing activities of daily living. The successful aging education component will cover topics including avoiding scams, fall prevention, living wills, and dementia awareness.
  Other Names: active control
  Arms: Successful Aging

SUMMARY:
The RAATE-MCI proposal is designed to determine the effects of physical activity on risk factors for Alzheimer's Disease in older African American adults. The study will compare a physical activity program to an active control group. RAATE-MCI is a 52-week randomized controlled trial. 144 African American adults aged 60 and older will be recruited.

DETAILED DESCRIPTION:
Regular physical activity has proven to be a safe and effective means to enhance cognitive function in older adults ranging from cognitively healthy to mildly cognitively impaired. A large body of existing data suggests that exercise improves cardiovascular and cerebrovascular functioning and thus has the potential to enhance perivascular clearance of amyloid and reduce chronic brain tissue ischemia, among other beneficial effects. Therefore, our study is focused on physical activity promotion, a potent approach to modifying multiple neurobiological pathways implicated in Alzheimer's Disease. RAATE-MCI is a 52-week randomized controlled trial that will assign insufficiently active African American adults aged 60 and older to one of two groups: a physical activity intervention or a successful aging (active control) group. Outcome measures will be collected at baseline, 24-,and 52-weeks. 144 older African American adults will be recruited.

Intervention will consist of one of two groups: a 150 minutes of physical activity (PA) per week or successful aging (SA) group. All physical activity and successful aging group sessions will be conducted at Pennington Biomedical or at local community facilities that include branches of the YMCA and community centers.

ELIGIBILITY:
Inclusion Criteria:

1. are African American (self-identify)
2. are 60 and older
3. are physically capable of exercise
4. are willing to accept randomization
5. are willing to attend group sessions
6. plan to live in the study area over the next 13 months and capable of traveling to designated study facility for clinic visits and intervention sessions for the next year
7. are free of conditions (e.g. uncontrolled asthma, severe sickle cell disease, etc.) that would make regular exercise unsafe as deemed by the medical investigator
8. have not engaged in regular physical activity
9. have a Short Physical Performance Battery ≥4
10. physically capable of exercise
11. are unable to utilize devices and/or applications as required for study participation
12. willing to attend group sessions
13. willing to allow researchers to use data for research purposes after study participation is completed
14. meet criteria for MCI as defined by the NIA-AA research framework a. cognitive performance below normal range (score < 1.5 SDs below the mean on NIH Toolbox scores for their age and sex on at least one of the subtests)

Exclusion Criteria:

1. have cognitive impairment that would interfere with participating in a group discussion

   a. cognitive performance in the demented range (score < 3 SDs below the mean on NIH Toolbox scores for their age and sex on at least one of the subtests)
2. meet criteria for dementia
3. are unwilling to give written informed consent or accept randomization in either study group
4. are too active (as defined by ≥10 min bouts of MVPA as measured by Actigraph) if:

   1. Sum of MVPA bouts for the 7 day wear period ≥40 mins
   2. Or ≤40 mins of MVPA 10min bouts AND ≥3 days of bouts
5. have uncontrolled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg).
6. have had a myocardial infarction, major heart surgery (i.e., valve replacement or bypass surgery), stroke, deep vein thrombosis, pulmonary embolus, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
7. are undergoing cardiopulmonary rehabilitation
8. have uncontrolled diabetes that in the judgment of the MI may interfere with study participation
9. have clinically diagnosed osteoporosis that in the judgment of the MI may interfere with study participation
10. are currently enrolled in another randomized trial involving lifestyle or pharmaceutical interventions
11. have another member of the household that is a participant in RAATE or RAATE MCI
12. refuse to participate in the study without disclosure of their amyloid PET scan results
13. refuse to allow anonymized versions of their study data for research after this study is completed.
14. have other medical, psychiatric, or behavioral factors that in the judgment of the Principal or Medical Investigator may interfere with study participation or the ability to follow the intervention protocol

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in executive function | Baseline, 24 weeks, 52 weeks
  The primary outcome measure will be executive function measured by the NIH-Toolbox Cognitive Battery. The NIH Toolbox Executive Function subdomain consists of the Flanker Inhibitory Control and Attention Test and the Dimensional Change Card Sort Test. The Flanker test is a measure of one's ability to inhibit attention to irrelevant conditions. Participants must identify the direction of a central visual stimuli amongst flanking stimuli either congruent or incongruent with the central stimuli. There are 40 trials and scores range from 0 - 10. The Card Sort is a measure of the ability to shift attention based on rules. Participants must match a target visual stimuli to either a color or word stimuli and this matching shifts during the assessment.
Change in episodic memory | Baseline, 24 weeks, 52 weeks
  The Rey Auditory Verbal Learning Test (RAVLT) is a common neuropsychological tool used to evaluate episodic memory. The RAVLT involves providing participants with 15 unrelated words and asking them to recall the word list. There are 5 trials designed to determine short-term memory and then a 30 minute delay to assess long-term memory. The total words correct in both the short- and long-term trials are used as outcome measures.

SECONDARY OUTCOMES:
Change in cognitive status | Baseline, 24 weeks, 52 weeks
  The Mini-Mental Status Examination is 30-point questionnaire to assess cognitive impairment.
Change in glucose | Baseline, 24 weeks, 52 weeks
  Fasting levels of glucose will be assessed using standard assays.
Change in time spent in physical activity | Baseline, 24 weeks, 52 weeks
  The Actigraph WGT3X+ accelerometer (ActiGraph LLC, Pensacola, FL) will be worn by the participant for a 7-day period. The device provides both the number of steps per day as well as time in sedentary, light, moderate, and vigorous activity in 1-minute epochs (for adults) using the default filter.
Change in cardiorespiratory fitness | Baseline, 24 weeks, 52 weeks
  All participants will perform a standardized graded exercise testing protocol administered on a treadmill. Fitness will be measured in terms of mL oxygen/kg/min.
Change in physical function-NIH Toolbox | Baseline, 24 weeks, 52 weeks
  Physical function will be assessed using the NIH-TB Motor assessment, which assesses dexterity, balance, locomotion, grip strength, and strength.
Change in telomere length | Baseline, 24 weeks, 52 weeks
  DNA will be extracted from the blood draw and amplified using real-time quantitative polymerase chain reaction (qPCR) to determine average relative telomere length represented by the telomere repeat copy number to single gene copy number (T/S) ratio in triplicate as previously described
Change in weight | Baseline, 24 weeks, 52 weeks
  Weight will be measured using a standard stadiometer. Measurements will be taken to the nearest cm.
Change in brain structure | Baseline, 24 weeks, 52 weeks
  Volumes of the cranial vault, brain tissue, gray matter, white matter, and cerebrospinal fluid, which will be provided as the primary brain structural outcome measures of interest from MRI.
Changes in brain function | Baseline, 24 weeks, 52 weeks
  Pre-selected inhibitory control ROIs (ACC for the Stroop; DLPFC, thalamus, superior frontal, inferior frontal, fusiform, and middle frontal gyri; and ACC and middle frontal gyri for the ANT) are of primary interest.
Change in lipoproteins | Baseline, 24 weeks, 52 weeks
  Fasting levels of lipids will be assessed using standard assays.
APOE genotype | Baseline
  APOE genotype will be assessed using standard assays.
Change in physical activity | Continuously for 52 weeks
  The Fitbit Charge 2 will be worn by participants in both groups.
Change in systolic blood pressure | SV, 26 weeks, 52 weeks
  Systolic blood pressure will be measured using the Omron, Model BP710 automatic blood pressure cuff.
Change in diastolic blood pressure | SV, 26 weeks, 52 weeks
  Diastolic blood pressure (both systolic and diastolic) will be measured using the Omron, Model BP710 automatic blood pressure cuff.
Change in mood | Baseline, 24 weeks, 52 weeks
  The Geriatric Depression Scale will be used to measure depressive symptoms.
Change in height | Baseline, 24 weeks, 52 weeks
  Height will be assessed using a standard stadiometer.
Change in physical function-SPPB | Baseline, 24 weeks, 52 weeks
  Physical function will be assessed using the the Short Physical Performance Battery (SPPB), which is a brief performance battery based on timed short distance walk, repeated chair stands and balance test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Newton, Jr., PhD, Principal Investigator — Pennington Biomedical Research; Owen Carmichael, PhD, Principal Investigator — Pennington Biomedical Research
Locations (1):
- Pennington Biomedical Research, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
For all study data, Pennington Biomedical has a well-structured internal process for data sharing and transfer. The Office of Legal and Regulatory Compliance is responsible for all data agreements which includes data subject to the protection under HIPAA. As part of the Louisiana State University System, Pennington Biomedical ensures that data agreements are in place in the following circumstances: business associate agreements when the transfer of data contains all identifiers, data use agreements when the transfer of data contains those identifiers that constitute a limited data set and a data transfer agreement in instances where data is de-identified, but still may be subject of protection in order to protect intellectual property rights. Transmission of data to ensure proper safeguards are in place on the data in motion and data at reset are carried out with assistance of the Research Computing Group or the Office of Computing Services.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after data analysis has occurred.